CLINICAL TRIAL: NCT05237661
Title: Study to Evaluate the Efficacy of Your Super's Moon Balance and Its Impact on Premenstrual Syndrome and Menstrual Symptoms
Brief Title: Study to Evaluate Your Super's Moon Balance and Its Impact on Premenstrual Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Your Super, INC. (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20230MoonBalance
Record Dates: First submitted 2022-02-02; First posted 2022-02-14 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: PMS; Menstrual Discomfort; Menstrual Pain
MeSH Terms: conditions — Dysmenorrhea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dietary supplement (Experimental): Dietary supplement: Moon Balance
  Interventions: Dietary Supplement: Moon Balance

INTERVENTIONS:
Dietary Supplement: Moon Balance — Moon Balance is a blend of 6 food ingredients

SUMMARY:
This is an open-label observational single-group clinical trial to study the efficacy of a commercially available dietary supplement and its effect on common PMS and menstrual symptoms, as well as health-related biomarkers.

DETAILED DESCRIPTION:
It is hypothesized that the dietary supplement marketed as "YOUR SUPER Moon Balance" will improve subjective wellbeing in trial participants by alleviating common symptoms of PMS and menstrual symptoms, such as pain, cramps, bloating, and lack of energy. Further, the ability of the supplement to reduce biomarkers of inflammation (CRP) and stress (cortisol), and promote sleep, will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with a regular menstruation
* Age 18-40
* Moderate self-reported discomfort during menstruation-related to bloating, cramps, fatigue, mood swings, or other PMS-related symptoms
* Must be in generally good health - no unstable, uncontrolled health condition
* BMI under 35
* Self-reported sleep-issues
* Willingness to refrain from ibuprofen or naproxen sodium (such as Advil, Aleve, Motrin or Midol) during each period (pill bleed) during the study
* Agree to not change their diet significantly during the duration of the study
* Agree to not change the intensity of their workouts for the duration of the study
* Must get their period regularly

Exclusion Criteria:

* Severe chronic conditions, including oncological and psychiatric disorders
* Known to have any severe allergic reactions
* Currently pregnant, breastfeeding, or wanting to become pregnant for the duration of the study
* Participants unwilling to follow the study protocol
* Have used a similar product (ingredients) in the 6 weeks prior to the study

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Gender identity
Enrollment: 38 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Change in perceived discomfort associated with menstruation | 12 weeks
  Perceived discomfort caused by several of the most common menstrual symptoms (energy, sleep, mood, comfort, and overall fewer PMS symptoms)
  Each endpoint will be reported by the participant on a scale of perceived discomfort at the end of each menstrual cycle. Participants will complete the surveys for each menstrual cycle. The study uses a questionnaire including a scale from 0-7 to assess the severity of symptoms(0=no symptoms and 7=very severe symptoms).

SECONDARY OUTCOMES:
Change in blood biomarkers: C-reactive protein | 12 weeks
  Change in C-Reactive Protein (CRP) with an at-home blood test after 12 weeks compared to baseline results.
Changes in saliva cortisol levels | 12 weeks
  Change in saliva cortisol levels with an at-home test after 12 weeks compared to baseline results.

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Mitschke, Principal Investigator — Citruslabs
Locations (1):
- Citruslabs, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: Undecided